CLINICAL TRIAL: NCT03032640
Title: Interactions of Human Gut Microbiota With Intestinal Sweet Taste Receptors
Acronym: ISTAR-micro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TRIMDFH 982524
Record Dates: First submitted 2016-11-11; First posted 2017-01-26 (Estimated); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Obesity
Keywords: Glucose; Sweet taste receptors; Artificial sweeteners
MeSH Terms: conditions — Obesity | interventions — Glucose Tolerance Test; Saccharin; lactisole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1- Healthy Lean subjects (Active Comparator): Group 1 will receive Sodium Saccharin 200mg capsule, 2x/day, Day 1-14
  Interventions: Other: Oral Glucose Tolerance Test (OGTT); Other: Assessment of dietary compliance; Other: Stool sampling; Other: Sodium Saccharin
- Group 2- Healthy Lean subjects (Active Comparator): Group 2 will receive Placebo 500mg capsule, 2x/day, Day 1-14
  Interventions: Other: Oral Glucose Tolerance Test (OGTT); Other: Assessment of dietary compliance; Other: Stool sampling; Other: Placebo
- Group 3- Healthy Lean subjects (Active Comparator): Group 3 will receive Sodium Saccharin 200mg + lactisole 335mg capsule, 2x/day, Day 1-14
  Interventions: Other: Oral Glucose Tolerance Test (OGTT); Other: Assessment of dietary compliance; Other: Stool sampling; Other: Sodium Saccharin; Other: Lactisole
- Group 4- Healthy Lean subjects (Active Comparator): Group 4 will receive Lactisole 335mg capsule, 2x/day, Day 1-14
  Interventions: Other: Oral Glucose Tolerance Test (OGTT); Other: Assessment of dietary compliance; Other: Stool sampling; Other: Lactisole

INTERVENTIONS:
Other: Oral Glucose Tolerance Test (OGTT) — Once we test the fasting plasma glucose (after an overnight fast), subject will receive a 75g glucose beverage they will have to drink within 5 minutes. Then after drinking the beverage, 8 blood samples will be collected through the IV catheter, over the next 3 hours.
Other: Assessment of dietary compliance — Assessment of consumption of non-caloric artificial sweeteners
Other: Stool sampling — Subjects will provide a stool sample.
Other: Sodium Saccharin — Subjects in group 1 and group 3 will be provided with sodium saccharin.
  Arms: Group 1- Healthy Lean subjects; Group 3- Healthy Lean subjects
Other: Placebo — Subjects in group 2 will be provided with placebo.
  Arms: Group 2- Healthy Lean subjects
Other: Lactisole — Subjects in group 3 and group 4 will be provided with lactisole.
  Arms: Group 3- Healthy Lean subjects; Group 4- Healthy Lean subjects

SUMMARY:
The purpose of this study is to collect data to examine whether short-term consumption of non-caloric artificial sweeteners (NCASs), such as saccharin, can lead to changes in blood sugar levels and in the composition of the bacteria in the large intestine.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent
2. Age 18-45 years
3. Weight stable (± 3 kg) during the 6 months prior to enrollment
4. BMI ≤ 25 kg/m2
5. Consumption of less than a can of diet beverage or a spoonful of NCASs weekly (or each equivalent from foods) during the past month

Exclusion Criteria:

1. Known coronary artery disease, angina or congestive heart failure
2. Type 1 or Type 2 Diabetes (A1c ≥6.5%)
3. Bleeding disorders
4. Hemoglobin level < 12.5 g/dL for women; hemoglobin level < 13.0 g/dL for men
5. Acute or chronic infections
6. Hepatitis and/or cirrhosis
7. Severe asthma or chronic obstructive pulmonary disease
8. Renal insufficiency or nephritis (creatinine > 1.6 mg/dl)
9. Prior bariatric surgery
10. Inflammatory bowel disease or malabsorption
11. Cancer within the last 3 years (except non-melanoma skin cancer or treated cervical carcinoma in situ)
12. Psychiatric disorders or eating disorders
13. Cushing's disease or syndrome
14. Untreated or inadequately controlled hypo- or hyperthyroidism (abnormal TSH)
15. Active rheumatoid arthritis or other inflammatory rheumatic disorder
16. Pregnant or nursing women
17. Smoking (smoking within the past 3 months)
18. Less than 4 bowel movements per week
19. Known hypersensitivity to saccharin, lactisole or any of its excipients.

    Excluded medications include but are not limited to:
20. Anti-diabetic agents
21. Oral, injected or chronic topical steroids (inhaled steroids for mild asthma are acceptable)
22. Antibiotic use (within the past 3 months)
23. Other drugs known to affect immune or metabolic function
24. Orlistat, phentermine, topiramate or other weight loss or anorectic agents (tricyclic antidepressants, atypical antipsychotics or other psychiatric drugs with effects on body weight)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Blood analyzed by way of NOVA StatStrip Meter and Milliplex Map Kit. | 6 weeks

SECONDARY OUTCOMES:
Short chain fatty acid analyses | 6 weeks
  Stool sample aliquoted and frozen by way of ribosomal sequencing, which will be used to determine what bacteria is in the fecal sample.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pratley, MD, Principal Investigator — Translational Research Institute for Metabolism and Diabetes
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swithers SE. Artificial sweeteners produce the counterintuitive effect of inducing metabolic derangements. Trends Endocrinol Metab. 2013 Sep;24(9):431-41. doi: 10.1016/j.tem.2013.05.005. Epub 2013 Jul 10. PMID 23850261
- [Background] Tilg H, Kaser A. Gut microbiome, obesity, and metabolic dysfunction. J Clin Invest. 2011 Jun;121(6):2126-32. doi: 10.1172/JCI58109. Epub 2011 Jun 1. PMID 21633181
- [Background] Suez J, Korem T, Zeevi D, Zilberman-Schapira G, Thaiss CA, Maza O, Israeli D, Zmora N, Gilad S, Weinberger A, Kuperman Y, Harmelin A, Kolodkin-Gal I, Shapiro H, Halpern Z, Segal E, Elinav E. Artificial sweeteners induce glucose intolerance by altering the gut microbiota. Nature. 2014 Oct 9;514(7521):181-6. doi: 10.1038/nature13793. Epub 2014 Sep 17. PMID 25231862
- [Background] Saccharin and its salts. IARC Monogr Eval Carcinog Risks Hum. 1999;73:517-624. No abstract available. PMID 10804968
- [Background] Pantarotto C, Salmona M, Garattini S. Plasma kinetics and urinary elimination of saccharin in man. Toxicol Lett. 1981 Dec;9(4):367-71. doi: 10.1016/0378-4274(81)90012-6. PMID 7330898
- [Background] Sweatman TW, Renwick AG. The tissue distribution and pharmacokinetics of saccharin in the rat. Toxicol Appl Pharmacol. 1980 Aug;55(1):18-31. doi: 10.1016/0041-008x(80)90215-x. No abstract available. PMID 7191585
- [Background] Renwick AG. The metabolism of intense sweeteners. Xenobiotica. 1986 Oct-Nov;16(10-11):1057-71. doi: 10.3109/00498258609038983. PMID 3541395
- [Background] Arnold DL, Krewski D, Munro IC. Saccharin: a toxicological and historical perspective. Toxicology. 1983 Jul-Aug;27(3-4):179-256. doi: 10.1016/0300-483x(83)90021-5. PMID 6353664
- [Background] Sweatman TW, Renwick AG, Burgess CD. The pharmacokinetics of saccharin in man. Xenobiotica. 1981 Aug;11(8):531-40. doi: 10.3109/00498258109045864. PMID 7303723
- [Background] Renwick AG. The disposition of saccharin in animals and man--a review. Food Chem Toxicol. 1985 Apr-May;23(4-5):429-35. doi: 10.1016/0278-6915(85)90136-x. PMID 3891556
- [Background] Evaluation of certain food additives and contaminants. Forty-first report of the Joint FAO/WHO Expert Committee on Food Additives. World Health Organ Tech Rep Ser. 1993;837:1-53. No abstract available. PMID 8266711
- [Background] Food and Agriculture Organization World Health Organization. Evaluation of certain food additives. Fifty-ninth report of the Joint FAO/WHO Expert Committee on Food Additives. World Health Organ Tech Rep Ser. 2002;913:i-viii, 1-153, back cover. PMID 12677645
- [Derived] Serrano J, Smith KR, Crouch AL, Sharma V, Yi F, Vargova V, LaMoia TE, Dupont LM, Serna V, Tang F, Gomes-Dias L, Blakeslee JJ, Hatzakis E, Peterson SN, Anderson M, Pratley RE, Kyriazis GA. High-dose saccharin supplementation does not induce gut microbiota changes or glucose intolerance in healthy humans and mice. Microbiome. 2021 Jan 12;9(1):11. doi: 10.1186/s40168-020-00976-w. PMID 33431052
- See also: Website for Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org